CLINICAL TRIAL: NCT03341455
Title: Developing, Implementing and Evaluating Preschool Based Interventions to Address Family Violence and Alcohol and Drug Misuse in Sri Lanka
Brief Title: Family Violence and Alcohol and Drug Misuse in Sri Lanka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Australian National University (Other)
Collaborators: University of Peradeniya (Other); Department of Foregin Affairs and Trade, Australia (Other Government)
Responsible Party: Principal Investigator, Polly Wallace, Co-investigator, Australian National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/066
Record Dates: First submitted 2017-04-12; First posted 2017-11-14 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Intimate Partner Violence; Domestic Abuse; Drug and Alcohol Abuse
Keywords: Sri Lanka; preschool; randomized control trial
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study will be implemented using a randomised controlled trial design. Parents with children attending government-managed preschools in two study areas will be recruited to participate. Preschools will be randomly assigned to an intervention or control group. Preschool teachers in the intervention group will also be recruited to participate.
Who Masked: Participant
Masking Description: Allocation of interventions cannot be concealed from either training staff or study participants once implementation occurs.
  All data collectors will be blinded to the intervention status of preschools.
  The study will be presented as a project related to family health and wellbeing, no specific study hypotheses will be presented to participants, and data collectors will not be involved in delivering the intervention. However, parents at preschools receiving the intervention will be aware of the training activities, and may still link the intervention to survey activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention preschools (Other): Capacity building to support families affected by IPV & substance misuse will be provided to the intervention preschools.
  Specifically, capacity building, training and support will be provided to
  * selected mothers on the provision of safe, confidential and relevant community-based referral and support services for women affected by IPV.
  * selected fathers on the provision of safe, confidential and relevant community-based referral and support to men seeking support for substance misuse problems.
  * intervention preschool teachers on provision of IPV and substance misuse prevention educational messages and referral pathways to services for these issues.
  Interventions: Behavioral: Capacity building to support families affected by IPV & substance misuse
- Control preschool (No Intervention): No intervention or training will not be provided to the control group in order to assess the impact of the intervention between the control and intervention arms of the study.

INTERVENTIONS:
Behavioral: Capacity building to support families affected by IPV & substance misuse — Training targeted groups (mothers, fathers, preschool teachers, community officers managing preschools) separately with the aim to identify and support high-risk families early enough to arrest the cycle of violence that results in children themselves becoming victims and perpetrators of such violence.
  Arms: Intervention preschools

SUMMARY:
The investigators aim to implement a community-based support program delivered by preschool teachers and volunteer parents that will increase awareness, knowledge and uptake of available services for IPV and substance misuse, and of the link between these issues and poorer education outcomes in children. Through this, the aim is to decrease the prevalence of IPV and substance misuse.

The proposed method of implementation is to deliver targeted training to preschool teachers, mothers with children at the preschools, fathers with children at the preschools, and community development officers managing preschools. This project will target the most vulnerable sections of the community and will provide a sustainable and feasible strategy for scale up of the intervention.

By intervening through these preschools the investigators aim to identify and support high-risk families early enough to arrest the cycle of violence that results in children themselves becoming victims and perpetrators of such violence.

DETAILED DESCRIPTION:
This project will be implemented as a cluster-randomised controlled trial (RCT) in preschools in 2 urban study areas. The unit of randomisation will be the preschool.

The intervention is a preschool-based capacity-building and support intervention addressing family violence and alcohol and drug misuse.

The study intervention will be delivered to preschool teachers, local government Community Development Department staff, other key government service providers, and selected mothers and fathers of children attending each preschool. Participants in data collection will be all teachers and parents of children in participating preschools.

Half the preschools in the study areas, selected at random, will receive the intervention initially. Those that do not will act as time-concurrent controls. If the intervention is demonstrated as being effective at the end of the study, these control preschools will subsequently receive the intervention.

This research will address important gaps in literature documented by other researchers by using multiple sources of data to assess the effectiveness of the intervention. Preschool communities have not previously been target populations when addressing domestic violence in Sri Lanka. Results will add to the evidence base for future interventions in Sri Lanka and have potential to contribute to national policy.

Study activities are listed in brief below, and will be subsequently expounded upon in the following sections.

1. A baseline survey at project outset will include mothers and fathers of children utilising these preschools, and will be conducted at the beginning of semester 1 of the project. This survey will include a series of self-report questionnaires, measuring: prevalence of family violence, prevalence of alcohol and drug misuse, depression, child psychological wellbeing, and gender attitudes to establish any baseline differences in prevalence of these factors between intervention and control groups.
2. Selected mothers and fathers from half of the preschools (the intervention group), along with preschool teachers, community development officers, and other government service providers, will receive training associated with the intervention before the end of semester 1.
3. Post intervention surveys with parents will be conducted near the end of the school year (at least 6 months post intervention) in all preschools in both study areas (both intervention and non-intervention groups).
4. Qualitative interviews will also be carried out with key informants associated with the project who received the intervention including teachers, community members, community development staff and other government sector service providers to determine their satisfaction with the intervention, and any challenges or barriers to its implementation.
5. If the intervention is deemed to have been effective, the non-intervention preschools will then receive the training intervention in 2019.

ELIGIBILITY:
Inclusion Criteria:

* parents must have at least one child attend the targeted preschool
* all participants must be literate in Tamil or Sinhalese or English

Exclusion Criteria:

- anyone with literacy difficulties (as the questionnaires are self-administered)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Difference in prevalence between the intervention and control groups of family violence experienced by preschool mothers. | At least six months post intervention
  Mothers from all participating preschools ( both intervention and control groups) will be surveyed to measure prevalence of family violence at 6 months after implementation of the intervention. The survey for mothers will include questions adapted from the World Health Organization Multi Country Survey of Violence against Women that will indicate prevalence of violence against them by their husband (or intimate partner). The survey will also include the Sri Lankan specific Peradeniya Depression Scale to measure mental health and depression in adults.

SECONDARY OUTCOMES:
Difference in prevalence between the intervention and control groups of alcohol and drug misuse experienced by preschool fathers. | At least six months post intervention
  Volunteer fathers from the preschool will be surveyed to measure the impact of the intervention on prevalence of alcohol and drug misuse. This survey will include locally validated versions of the Alcohol Used Disorders Identification Test (AUDIT), the Drug Abuse Screening Test (DAST) and the Sri Lankan specific Peradeniya Depression Scale to measure mental health and depression in adults.

CONTACTS AND LOCATIONS:
Overall Officials: Kamalini Lokuge, Dr, Principal Investigator — Humanitarian Research Project Leader
Locations (1):
- Australian National University, Canberra, Australian Capital Territory, Australia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Derived] Lokuge K, Wallace P, Subasinghe K, Thurber K, De Silva T, Clarke N, Waas D, Liyanage N, Attygalle U, Carron-Arthur B, Rodrigo K, Banks E, D'Este C, Rajapakse T. Protocol for a cluster-randomised controlled trial evaluating the impact of a preschool-based capacity building intervention on intimate partner violence and substance misuse in Sri Lanka. BMC Public Health. 2018 May 2;18(1):572. doi: 10.1186/s12889-018-5423-8. PMID 29716553